CLINICAL TRIAL: NCT03904459
Title: The Norwegian JIA Study - Temporo-mandibular Involvement, Oral Health, Uveitis, Bone Health and Quality of Life in Children With Juvenile Idiopathic Arthritis (JIA). A Large Multicentre Study
Brief Title: Jaw, Mouth and Bone Health, and Quality of Life in Children With Juvenile Idiopathic Arthritis (JIA)
Acronym: NorJIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: St. Olavs Hospital (Other); University Hospital of North Norway (Other); Oral Health Centre of Expertise Mid, North and West Norway (Unknown); Norwegian University of Science and Technology (Other); University of Tromso (Other); University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: NorJIA
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Arthritis, Juvenile
Keywords: Temporomandibular Joint; Oral Health; Bone & Bones; Bone Density; Quality of Life
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, stimulated and unstimulated saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: Children with juvenile idiopathic arthritis
  Interventions: Other: no intervention
- controls: healthy children
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The Norwegian JIA Study (NorJIA) is a prospective, longitudinal, multicenter, observational study of 250 children with juvenile idiopathic arthritis (JIA) and 250 healthy controls, attending the three Norwegian university clinics in Bergen, Tromsø, or Trondheim. The study will run over 5 years, and include extensive clinical, laboratory, radiological and oral examinations at baseline and after 2 years follow-up. There will be a special focus on the jaw (temporomandibular joints) with extensive imaging and clinical examination, aiming at establishing scoring systems for active and chronic disease and growth disturbances. Another focus is to study mouth and teeth problems, such as caries and gingivitis, and look for predictors of poor oral health in children with JIA compared to health peers. As chronic inflammation, reduced physical activity and certain anti-inflammatory drugs can be detrimental for bone strength and development, the investigators also want to study the bone health of children with JIA, and look for predictors of poor bone mineral density. The results of the study may contribute to better diagnostics of inflammatory processes, earlier detection of poor oral or bone health, and thereby point to possible prevention strategies to increase quality of life for children with JIA in the future.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the ILAR criteria for juvenile idiopathic arthritis

Exclusion Criteria:

* no consent

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with juvenile idiopathic arthritis followed at any of the three participating centers according to hospital files. Controls are recruited at The Oral Health Centre of Expertise (Tk) Mid-Norway (TkMN), TkWest or at Tk Northern Norway (TkNN) from their lists of children due for a free visit to the dentist according to the Norwegian public dental service policy.
Sampling Method: Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 2 years
  measured by a Dual-energy X-ray absorptiometry (DXA) scan of the hip, lumbar spine and total body with body composition and expressed in Z scores, number of standard deviations (SD) from the expected mean according to sex and age
Joint inflammation and damage | 2 years
  defined according to predefined standard protocol for 3-Tesla MRI of the temporomandibular joints
caries experience DMFTS/dmfts | 2 years
  Measured by: DMFTS = Number of decayed/missed/filled permanent teeth in the age group 12-17 years, or dmfts = No. of decayed/missed/filled primary teeth in children up to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Ansgar Berg, Study Director — Department of Pediatrics, Haukeland University Hospital
Locations (5):
- Norway (5):
  - Oral Health Centre of Expertise West Norway, Bergen
  - Oral Health Centre of Expertise North Norway, Tromsø
  - University Hospital in North Norway, Tromsø
  - Oral heath Centre of Expertise Mid Norway, Trondheim
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundestad A, Cetrelli L, Angenete OW, Augdal TA, Tylleskar K, Nordal EB, Rosendahl K, Hoftun GB, Hoff M, Romundstad PR, Rygg M. Bone health in juvenile idiopathic arthritis compared with controls based on a Norwegian observational study. RMD Open. 2025 Jun 19;11(2):e005605. doi: 10.1136/rmdopen-2025-005605. PMID 40537274
- [Derived] Arneng SM, Jenssen IP, Lundestad A, Cetrelli L, Angenete O, Nordal E, Tylleskar KB, Romundstad PR, Rygg M. The patient's voice: a cross-sectional study of physical health and disability in juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2024 Nov 18;22(1):100. doi: 10.1186/s12969-024-01034-7. PMID 39558411
- [Derived] Halbig JM, Jonsson B, Gil EG, Astrom AN, Rypdal V, Frid P, Augdal TA, Fischer J, Cetrelli L, Rygg M, Lundestad A, Tylleskar K, Nordal E; Norwegian JIA Study - Temporo-mandibular Involvement, Oral Health, Uveitis, Bone Health, Quality of Life in Children with Juvenile Idiopathic Arthritis. Oral health-related quality of life, impaired physical health and orofacial pain in children and adolescents with juvenile idiopathic arthritis - a prospective multicenter cohort study. BMC Oral Health. 2023 Nov 20;23(1):895. doi: 10.1186/s12903-023-03510-0. PMID 37986155
- [Derived] Augdal TA, Angenete OW, Shi XQ, Sall M, Fischer JM, Nordal E, Rosendahl K. Cone beam computed tomography in the assessment of TMJ deformity in children with JIA: repeatability of a novel scoring system. BMC Oral Health. 2023 Jan 10;23(1):12. doi: 10.1186/s12903-022-02701-5. PMID 36627622
- [Derived] Fischer J, Skeie MS, Rosendahl K, Tylleskar K, Lie S, Shi XQ, Gil EG, Cetrelli L, Halbig J, von Wangenheim Marti L, Rygg M, Frid P, Stoustrup P, Rosen A. Prevalence of temporomandibular disorder in children and adolescents with juvenile idiopathic arthritis - a Norwegian cross- sectional multicentre study. BMC Oral Health. 2020 Oct 13;20(1):282. doi: 10.1186/s12903-020-01234-z. PMID 33050890
- See also: Related Info — http://www.norjia.com